CLINICAL TRIAL: NCT06841146
Title: Prediction of Adhesion by Sliding Sign in Three or Above Cesarean Section
Brief Title: Prediction of Adhesion by Sliding Sign
Acronym: Prediction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Alev Esercan, Sanliurfa Education and Research Hospital, Sanliurfa Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ŞEAH/CS
Record Dates: First submitted 2024-12-27; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adhesions Abdominal
Keywords: adhesion; cesarean section; sliding sign
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients that had cesarean section (Active Comparator): patients had ultrasonograpy done before cesarean section and sliding sign will be defined,and at cesarean section adhesions will be defined.
  Interventions: Procedure: routine cesarean section

INTERVENTIONS:
Procedure: routine cesarean section — cesarean section

SUMMARY:
Sliding sign will be checked by ultrasonography by transabdominal and transvaginal route before operation of patients that had cesarean section three or more. During cesarean section adhesions will be evaluated and noted. The correlation and predictive values of adhesion and sliding sign will be defined in our study.

DETAILED DESCRIPTION:
Three or more cesarean section patients will be included in our study. In addition, inflammatory markers in complete blood count as neutrophil, lymphocyte, neutrophil/ lymphocyte ratio, pan immune inflammation value (PIV) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* all three and above number of cesarean section patients

Exclusion Criteria: placenta adhesion spectrum

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-02-19 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
predictive value of sliding sign for adhesions intraabdominally | before cesarean section
  sensivitivity and specivitivity of sliding sign

IPD SHARING:
Plan to Share IPD: No